CLINICAL TRIAL: NCT03050853
Title: The Appeal and Impact of E-cigarettes in Smokers With Serious Mental Illness
Brief Title: The Appeal and Impact of E-cigarettes in Smokers With SMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Vinfen (Industry); Centerstone Kentucky (Unknown)
Responsible Party: Principal Investigator, Sarah Pratt, Scientist, Psych Research, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 29154
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Tobacco Dependence; Schizophrenia; Bipolar Disorder; Schizoaffective Disorder
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia; Bipolar Disorder; Psychotic Disorders | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: This is a study to learn about the appeal and health impacts of using e-cigarettes in people with serious mental illness who are not currently thinking about qutting smoking. Reduction of craving or quitting are not targets
Who Masked: Outcomes Assessor
Masking Description: All follow-up assessments will be conducted by the masked outcome assessor with the exception of the tobacco use and e-cigarette use self report and the satisfaction with e-cigarettes scale administered to the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-Cigarette (Experimental): The E-cigarette arm will be asked to use e-cigarettes in place of regular tobacco products. The group will be assessed at baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 13 weeks, and 26 weeks.
  Interventions: Behavioral: E-cigarette
- Assessments only (No Intervention): The Assessment only group will be asked to refrain from use of e-cigarettes during participation. The group will be assessed at baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 13 weeks, and 26 weeks.

INTERVENTIONS:
Behavioral: E-cigarette — The e-cigarette arm will be provided with 8 weeks of free e-cigarettes based on self-report of regular tobacco use. Participants assigned in this arm will be asked to switch combustible tobacco with e-cigarettes. The appeal of e-cigarettes and health impacts will be measured, but we are not targeting quitting combustible tobacco or reducing craving.
  Arms: E-Cigarette

SUMMARY:
This study will evaluate behavioral and psychological appeal, toxicity, and effect of e-cigarettes on smoking behavior and nicotine addiction in chronic smokers with serious mental illness (SMI) who have failed to quit smoking. A total of 240 participants will be enrolled and randomly assigned to either receive a supply of e-cigarettes for 8 weeks plus assessments (baseline & weeks 2, 4, 6, 8, 13, & 26) or assessments only. This single-blinded study will provide e-cigarettes and instructions on their safe use. Level of appeal will be inferred from carefully assessed use of e-cigarettes and reduction in combustible tobacco. Qualitative data will also be collected from participants assigned to e-cigarettes, given that unanticipated issues will almost certainly arise in connection with e-cigarette use that can only be captured within a qualitative debriefing at the conclusion of participants' time in the study.

DETAILED DESCRIPTION:
The main addictive component in tobacco, nicotine, has very low toxicity in cigarette doses and is available in a novel product, electronic cigarettes (e-cigarettes). E-cigarettes are widely available and popular; almost one-third of cigarette smokers in the general population have tried them. E-cigarette use may be equally common among heavily dependent subgroups of chronic smokers. For example, two studies suggest that smokers with mental illness have tried this product at similar or even higher rates compared with the general population. This proposal targets chronic, highly dependent smokers with serious mental illness (SMI) who have been unable to quit and are thus maintaining exposure to toxins in combustible tobacco smoke. Whether smokers with SMI find e-cigarettes appealing is an important question because substituting e-cigarettes for combustible cigarettes may have profound health effects related to reduced impact on lung function and cardiovascular inflammation, as well as reduced exposure to carcinogens and tumor promoters.

E-Cigarettes are popular and readily available even though information about toxicity, addiction liability, effect on health, and impact on current or future smoking behaviors is limited. Given the ubiquity of e-cigarette use and the lack of definitive data on their impact, more information about their appeal and impact, especially in vulnerable populations who are unable to quit smoking, will be key for regulators and treatment providers. The FDA has published its intention to regulate e-cigarettes, and the National Institute on Drug Abuse (NIDA) is supporting the development of a standardized, safety-tested e-cigarette for use in research. The American Heart Association recently issued a policy statement that e-cigarettes present "an opportunity for harm reduction if smokers adopt this alternative tobacco product as a substitute for cigarettes," but further research on behavioral and psychological appeal, toxicity, and impact of e-cigarettes on smoking heavier and nicotine dependence are sorely needed. The proposed study would add significantly to this science base.

In partnership with the New Hampshire Department of Medicaid, this research group conducted a statewide study of incentives for health behavior change. Over 600 smokers with mental illness were enrolled and randomly assigned to 1 of 3 smoking cessation treatments. Almost 23% of smokers with schizophrenia and 31% of smokers with bipolar disorder had tried an e-cigarette during the 3 months prior to participating in the study, providing evidence for the potential appeal of e-cigarettes among people with SMI who are trying to quit smoking.

These findings led to a preliminary prospective study of e-cigarette use among 19 chronic smokers (9 had bipolar disorder, 10 had schizophrenia) who had tried to quit an average of 3.8 (±8.14) times over the prior year but were no longer seeking cessation treatment. Participants received a 4-week supply of e-cigarettes and instruction on their safe use, and were assessed weekly for a month. Participants sustained a steady level of e-cigarette use over the study period. Overall, participants significantly reduced the number of cigarettes smoked per week from a mean of 191.9 (±159.3) at baseline to 66.7 (±76.3) at the final study visit (t=3.26, df=17, p=.005), confirmed by a significant decrease in mean CO level from 27ppm (±16.9) to 15ppm (±9.2) (t=3.246, df=18, p=.004). Participants rated several aspects of e-cigarette use based on items created for this study, including: 1) enjoyment compared to tobacco cigarettes, 2) satisfaction from e-cigarettes, and 3) willingness to buy e-cigarettes. Ratings were consistently high (>4 on a 5-point Likert type scale) across the 4 weeks. This study provides the basis and justification for conducting a large study using a randomized design to learn more about the behavioral and psychological appeal of e-cigarettes among chronic smokers with SMI, and to explore important aspects of e-cigarette use, including impact on toxicity and nicotine dependence.

This study will evaluate the behavioral and psychological appeal of e-cigarettes among chronic smokers with SMI, it will evaluate the effect of e-cigarettes on markers of tobacco toxicity, and it will evaluate the effect of e-cigarettes on measures of nicotine dependence. A total of 240 people with SMI who are receiving services at 1 of 2 mental health providers (Vinfen Corporation in Lowell/Lawrence MA and Centerstone Kentucky, formerly Seven Counties Services, Inc. in Louisville, KY) will be enrolled and randomly assigned.

The hypothesis is that at least 50% of smokers assigned to the e-cigarette group will use e-cigarettes daily during each of the 8 weeks that they are provided; mean satisfaction of e-cigarettes will be >3 on a 5-point scale; and subjective perception of e-cigarettes will be positive based on responses to a qualitative interview.

Secondly, it is hypothesized that over 8 weeks, reduction in expired breath CO, combustible cigarettes consumed/week, and urine levels of 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol or NNAL (a tobacco-specific carcinogen) will be greater among those assigned to e-cigarettes compared to those assigned to assessment only. Lastly, it is hypothesized that people assigned to e-cigarettes will have similar nicotine dependence at the end of the study period, when compared to people assigned to assessment only.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia, Schizoaffective Disorder, or Bipolar Disorder
* Enrolled in services at the research site for a minimum of 3 months
* Regular smoker (approximately 10 cigarettes for the past 5 years) with a history of at least 1 quit attempt
* Fluent in English

Exclusion Criteria:

* Regular use of e-cigarettes in the past month
* Current interest/plan to quit smoking
* Regular use of nicotine replacement therapy to quit smoking or use of bupropion or varenicline to quit smoking
* Use of emergency room or hospitalization for psychiatric reasons in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Carbon Monoxide Level | Baseline, 2 week, 4 week, 6 week, 8 week, 13 week, 26 week
  Carbon Monoxide Measurement
Change in Cancer Related Toxin, 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol or NNAL | Baseline, 4 week, 8 week, 13 week, 26 week
  Urine NNAL analysis
Change in the use of e-cigarettes | Baseline, 2 week, 4 week, 6 week, 8 week, 13 week, 26 week
  Count of e-cigarettes

SECONDARY OUTCOMES:
Change in Nicotine Dependence | Baseline, 2 week, 4 week, 6 week, 8 week, 13 week, 26 week
  Fagerstrom Test of Nicotine Dependence

CONTACTS AND LOCATIONS:
Overall Officials: Sarah I Pratt, Ph.D., Principal Investigator — Dartmouth College
Locations (2):
- United States (2):
  - Centerstone Kentucky, Louisville, Kentucky
  - Vinfen Corp, Lawrence, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benowitz NL. Clinical pharmacology of nicotine: implications for understanding, preventing, and treating tobacco addiction. Clin Pharmacol Ther. 2008 Apr;83(4):531-41. doi: 10.1038/clpt.2008.3. Epub 2008 Feb 27. PMID 18305452
- [Background] Polosa R, Rodu B, Caponnetto P, Maglia M, Raciti C. A fresh look at tobacco harm reduction: the case for the electronic cigarette. Harm Reduct J. 2013 Oct 4;10:19. doi: 10.1186/1477-7517-10-19. PMID 24090432
- [Background] Etter JF, Bullen C. Electronic cigarette: users profile, utilization, satisfaction and perceived efficacy. Addiction. 2011 Nov;106(11):2017-28. doi: 10.1111/j.1360-0443.2011.03505.x. Epub 2011 Jul 27. PMID 21592253
- [Background] Pratt SI, Sargent J, Daniels L, Santos MM, Brunette M. Appeal of electronic cigarettes in smokers with serious mental illness. Addict Behav. 2016 Aug;59:30-4. doi: 10.1016/j.addbeh.2016.03.009. Epub 2016 Mar 19. PMID 27043170
- [Derived] Sargent JD, Pratt SI, Brunette MF, Ferron JC, Santos MM, Stoolmiller M. Level and timing of product substitution in a trial of e-cigarettes for smokers not interested in quitting. Tob Induc Dis. 2024 Jun 13;22. doi: 10.18332/tid/189220. eCollection 2024. PMID 38873183
- [Derived] Pratt SI, Ferron JC, Brunette MF, Santos M, Sargent J, Xie H. E-Cigarette Provision to Promote Switching in Cigarette Smokers With Serious Mental Illness-A Randomized Trial. Nicotine Tob Res. 2022 Aug 6;24(9):1405-1412. doi: 10.1093/ntr/ntac082. PMID 35363874